CLINICAL TRIAL: NCT02329522
Title: Non-Invasive Doppler Ultrasound For Assessing Patients With Chronic Obstructive Pulmonary Disease: A Prospective Observational Study
Brief Title: USCOM For Assessing Patients With COPD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Timothy H Rainer, Director & Professor, Chinese University of Hong Kong
Other Study IDs: 2013.640
Record Dates: First submitted 2014-12-22; First posted 2014-12-31 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Haemodynamics; Chronic obstructive pulmonary disease; Ultrasonic Cardiac Output Monitor; severity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Spirometry; Respiratory Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Stable COPD patients: Patients will be assessed using USCOM and spirometry. For those with FEV1 to FVC ratio smaller than 70%, they will be classified as COPD.
  Interventions: Device: Ultrasonic Cardiac Output Monitor; Device: Spirometry
- AECOPD patients: Patients will be assessed using USCOM and spirometry. Spirometry will be assessed after 2 to 4 weeks post-hospital discharge.
  Interventions: Device: Ultrasonic Cardiac Output Monitor; Device: Spirometry
- Patient Controls: Patients will be assessed using USCOM and spirometry. For those with COPD symptoms but FEV1 to FVC ratio greater than 70%, they will be classified as non-COPD.
  Interventions: Device: Ultrasonic Cardiac Output Monitor; Device: Spirometry
- Healthy Controls: Healthy subjects, with no history of COPD or other significant chronic illness will be recruited as healthy controls. Subjects will be matched for age and gender with the patient groups. They will be assessed using USCOM.
  Interventions: Device: Ultrasonic Cardiac Output Monitor

INTERVENTIONS:
Device: Ultrasonic Cardiac Output Monitor — An Ultrasonic Cardiac Output Monitor (USCOM; USCOM Pty Ltd, NSW, Australia) is a non-invasive Doppler ultrasonography. It is capable of measuring haemodynamic parameters non-invasively and appears to be simple and rapid to use, portable, relatively inexpensive and has less potential complications compared with the standard technique, pulmonary artery thermodilution (PATD).
  USCOM scans will be performed on patients to measure direct and derived haemodynamic variables, which will be performed in the supine position wherever possible. A transducer will be placed on the chest in either the suprasternal position to measure trans-aortic blood flow, or the left parasternal position to measure transpulmonary blood flow.
  Other Names: USCOM
Device: Spirometry — Spirometry assesses lung function through measuring the amount (volume) and/or speed (flow) of air that can be inhaled and exhaled. Patients are regarded as COPD if their Forced expiratory volume in 1 second (FEV1) to Forced vital capacity (FVC) ratio are smaller than 70%. Patients were required to perform three blowing manoeuvres, and post-bronchodilator test results were obtained within 20 minutes to 4 hours after inhaling 400 mg of salbultamol.
  Other Names: Lung function test
  Groups: AECOPD patients; Patient Controls; Stable COPD patients

SUMMARY:
Objective

The Ultrasonic Cardiac Output Monitor (USCOM) is a non-invasive, quantitative method for measuring and monitoring cardiovascular haemodynamic parameters in patients. The aims of this study are:

1. To investigate whether there is any correlation between haemodynamic parameters and COPD severity.
2. To investigate whether USCOM-derived haemodynamic variables may be used as prognostic indicators of 6-month, 1-year, 3-year and 5-year readmission.
3. To investigate whether USCOM-derived haemodynamic variables may be used as prognostic indicators of 6-month, 1-year, 3-year and 5-year all-cause mortality.

Design, Setting and Subjects This prospective observational study will be conducted in the Prince of Wales Hospital in Hong Kong.

Interventions Haemodynamic measurements made using the USCOM, and spirometry, will be performed as appropriate on subjects in respiratory clinic, the emergency department, medical wards and on ICU. In order to assess inter-observer variability, a second, blinded operator will repeated 15% of scans.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is the fourth leading cause of death in the world, a lung disorder which is characterized by a partially reversible airflow limitation, which is usually progressive, and associated with an abnormal inflammatory response to noxious particles or gases. In 2005, among elderly Hong Kong Chinese (age ≥60 years) in Hong Kong with COPD defined as an FEV1/FVC <70%, 19.6% males and 11.9% females suffered from moderate levels of severity.

From an initial stable condition, an acute exacerbation of COPD (AECOPD) is characterized by a sudden onset of breathlessness, purulent sputum, and increases in sputum volume. Other symptoms include increasing cough, wheeze, chest tightness or fatigue. The major cause of AECOPD is infection, although other stimulating factors include air pollution, withdrawal of medication, and low temperature. After the first admission of an exacerbation, the readmission rate for patients with AECOPD is high. The mean number of annual readmissions is 2.2 episodes, with a one-year mortality rate of 14%.

Spirometry can help to diagnose COPD patients, and a post-bronchodilator FEV1/FVC<0.7 confirms the presence of airflow limitation. The classification of severity of airflow limitation in COPD is based on GOLD category. The lower the post-bronchodilator FEV1, the higher is the severity. This method is useful for assessing patients with stable COPD only. For those with AECOPD, this method may not be easy to conduct and assess patients immediately due to patients' difficulty in breathing.

A common dilemma facing clinicians is whether patients presenting with breathlessness, cough and wheeze have an acute exacerbation of COPD, an acute exacerbation of left ventricular failure (LVF), or some degree of both. Making an accurate diagnosis is important as the treatment in each case is different, and a quick recovery depends upon appropriate and timely intervention and treatment.

Unlike acute exacerbations of asthma, there are no objective guidelines on how to assess the severity and prognosis of patients presenting to hospital with acute exacerbations of COPD. However, the CURB65, originally intended for assessing patients with pneumonia, has been evaluated in this context. High CURB65 scores in patients presenting with acute exacerbations of COPD do predict increasing risk of hospital and one month mortality from 2 to 21% but do not predict patients with very high risk.

In healthy subjects, the presence or absence of carbon dioxide retention influences the body's haemodynamic response. Hypercapnia has been shown to increase mean pulmonary artery pressure (PAP), pulmonary vascular resistance (PVR), heart rate (HR), stroke volume (SV), cardiac output (CO), and mean arterial BP (MAP). However, hypercapnia does not appear to affect indices of systolic function, such as peak aortic velocity and aortic mean and peak acceleration, or plasma renin, angiotensin II, and aldosterone activity.

In stable patients with compensated COPD, elevations in CO2 trigger central and peripheral chemoreceptors resulting in an increased depth and rate of respiration, bradycardia (via vagal stimulation), and systemic vasoconstriction (via sympathetic stimulation). Therefore, cardiovascular parameters may be either normal or, if there is a degree of carbon dioxide retention resulting in catecholamine release and autonomic stimulation, then moderately hyperdynamic. Patients with COPD should have a cardiac Index (CI), which is elevated either towards the upper half or above the normal range, and may be as high as 5L/min/m2, an elevated SI, an elevated SVR and elevated DO2.

The Smith-Madigan Index II (SMII) is a novel measure of inotropy, which in stable COPD patients should either be normal or, if there are adrenergic effects, then may be elevated to as much as 1.6. The effects of hypercapnia in patients with COPD on potential to kinetic energy ratio (PE/KE, PKR), flow time (FT), peak velocity (Vpk) and mean pressure gradient (Pmn) are unknown.

These changes contrast with patients with acute LVF, where CI is low and the SMII is usually less than 1.0, and commonly around 0.7 - 0.8. PE/KE and SVR are generally much higher, and FT (as a function of SV) is longer. Vpk and Pmn are also lower in LVF.

We have conducted a preliminary study to evaluate the correlation between severity of COPD and haemodynamic parameters. 86 stable COPD patients, 43 AECOPD patients and 36 healthy, age and gender matched subjects were recruited. It was found that the severity of COPD correlated positively with mean heart rate, cardiac index (CI), ejection time percentage (ET%) oxygen delivery index (DO2I) and inotropy. When compared with healthy controls, stable GOLD IV patients had a significantly higher CI (3.98 vs 3.15 l/min/m2, p<0.005), inotropy (2.14 vs 1.72 W/m2, p<0.01) and DO2I (679.8 vs 530.7 ml/min/m2, p<0.01), and a significantly lower potential to kinetic energy ratio (PKR) (43.0 vs 56.6, p<0.05). Moreover, the 30-day readmission rate was the highest in GOPD IV patients. Based on the existing findings, it would be interesting to study the long-term prognostic effect of haemodynamic parameters in COPD patients.

Aim

The aims of the present study for patients visited respiratory clinic or admitted to the Emergency Department (ED), including those admitted to resuscitation room or emergency high dependency unit, are:

1. To investigate whether there is any correlation between haemodynamic parameters and COPD severity.
2. To investigate whether USCOM-derived haemodynamic variables may be used as prognostic indicators of 6-month, 1-year, 3-year and 5-year readmission.
3. To investigate whether USCOM-derived haemodynamic variables may be used as prognostic indicators of 6-month, 1-year, 3-year and 5-year all-cause mortality.

Measurements

* Haemodynamic measurements using an Ultrasonic Cardiac Output Monitor (USCOM®; USCOM Pty Ltd, NSW, Australia)
* Lung function assessment using Spirometry (MICROLAB 3300 spirometer; Micro Medical, Kent, UK)
* 6-minute walk test
* Borg dyspnoea scale
* Blood pressure
* End-tidal CO2

Definition of haemodynamic parameters:

* Velocity time integral (vti) is the integral of the flow profile, i.e. the distance the blood travels in one beat. The unit of vti is m/s.
* Cardiac output (CO) is the volume of blood pumped by the heart in one minute: CO = SV x HR. The unit is l/min.
* Cardiac index (CI) is equal to CO divided by BSA. The unit is l/min/m2.
* Stroke volume (SV) is the volume of blood ejected from the heart during one systolic stroke. SV = vti x πr2,where πr2 = flow cross sectional area. The unit of SV is ml.
* Stroke volume index (SVI) is SV divided by BSA and the unit is ml/m2.
* Stroke volume variation (SVV) is the percentage change in SV between a group of beats. SVV = (SVmax - SVmin x 100) / [(SVmax + SVmin)/2].
* Systemic vascular resistance (SVR) is the pressure against which the heart pumps. SVR = MAP/CO. The unit is d.s.cm-5.
* Systemic vascular resistance index (SVRI) SVRI = SVR x BSA d.s.cm-5m2.
* Oxygen delivery (DO2) is calculated by the equation: DO2 = 1.34 x Hb x SpO2/100 x CO, where Hb = hemoglobin in grams of hemoglobin per litre of blood (g/l); SpO2 = the peripheral oxygen saturation as a percentage (%). The unit of DO2 is ml/min.
* Oxygen delivery index (DO2I) is equal to DO2 divided by BSA. The unit of DO2I is ml/min/m2.
* Inotropy index refers to (Potential energy + Kinetic energy) divided by body surface area. The unit of inotropy is W/m2.
* Potential to kinetic energy ratio (PKR) is the energy used to produce blood pressure divided by the energy used to produce blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Age >40 years;
* Clinically diagnosed as COPD by physicians;
* Obtain any one of exacerbating symptoms (increased dyspnoea, sputum production, sputum volume, wheeze, cough or exertional dyspnoea);

Exclusion Criteria:

* Known or suspected pregnancy, lactating patients, active malignancies, severe mobility problems (e.g. significant painful arthritis), and confusion or dementia .

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a de novo diagnosis of COPD or a known history of COPD who attend a respiratory clinic or the emergency department in the Prince of Wales Hospital (Shatin, Hong Kong) will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-10 (Actual); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
The difference in mean cardiac index (CI) among the Global Initiative for Chronic Obstructive Lung Disease (GOLD) stage I, II, III, IV and healthy subjects. | On Day 1

SECONDARY OUTCOMES:
The difference in velocity time interval (vti) obtained using USCOM among GOLD stage I, II, III, IV and healthy subjects | On Day 1
  USCOM - Ultrasonic Cardiac Output Monitor Please see the definition of the haemodynamic parameters in Detailed Description.
The differences in USCOM-derived haemodynamic parameters, including CO, SV, SVI, SVV, SVR, SVRI, DO2, DO2I, Intropy and PKR obtained using USCOM among GOLD stage I, II, III, IV and healthy subjects | On Day 1
  Please see the definition of the haemodynamic parameters in Detailed Description.
  Abbreviation: cardiac output (CO), stroke volume (SV), stroke volume index (SVI), stroke volume variation (SVV), systemic vascular resistance (SVR), systemic vascular resistance index (SVRI), oxygen delivery (DO2), oxygen delivery index (DO2I), Intropy and potential to kinetic energy ratio (PKR)
The differences in USCOM-derived haemodynamic parameters, including CO, CI, SVR, SVRI, SVV, DO2, DO2I, Intropy and PKR between stable and acute exacerbated condition | On Day 1
  Please see the definition of the haemodynamic parameters in Detailed Description.
  Abbreviation: cardiac output (CO), cardiac index (CI), systemic vascular resistance (SVR), systemic vascular resistance index (SVRI), stoke volume variation (SVV), oxygen delivery (DO2), oxygen delivery index (DO2I), Intropy and potential to kinetic energy ratio (PKR).
The number of 6-month, 1-year, 3-year and 5-year readmission in COPD patients | Year 5
The number of 6-month, 1-year, 3-year and 5-year all-cause mortality in COPD patients | Year 5

CONTACTS AND LOCATIONS:
Overall Officials: Timothy H Rainer, MD FCEM, Principal Investigator — Accident & Emergency Medicine Academic Unit
Locations (1):
- Prince of Wales Hospital, Hong Kong, China

REFERENCES:
- [Background] Ko FW, Woo J, Tam W, Lai CK, Ngai J, Kwok T, Hui DS. Prevalence and risk factors of airflow obstruction in an elderly Chinese population. Eur Respir J. 2008 Dec;32(6):1472-8. doi: 10.1183/09031936.00058708. Epub 2008 Aug 6. PMID 18684847
- [Background] Wedzicha JA. Role of viruses in exacerbations of chronic obstructive pulmonary disease. Proc Am Thorac Soc. 2004;1(2):115-20. doi: 10.1513/pats.2306030. PMID 16113423
- [Background] Anderson HR, Spix C, Medina S, Schouten JP, Castellsague J, Rossi G, Zmirou D, Touloumi G, Wojtyniak B, Ponka A, Bacharova L, Schwartz J, Katsouyanni K. Air pollution and daily admissions for chronic obstructive pulmonary disease in 6 European cities: results from the APHEA project. Eur Respir J. 1997 May;10(5):1064-71. doi: 10.1183/09031936.97.10051064. PMID 9163648
- [Background] Wouters EF, Postma DS, Fokkens B, Hop WC, Prins J, Kuipers AF, Pasma HR, Hensing CA, Creutzberg EC; COSMIC (COPD and Seretide: a Multi-Center Intervention and Characterization) Study Group. Withdrawal of fluticasone propionate from combined salmeterol/fluticasone treatment in patients with COPD causes immediate and sustained disease deterioration: a randomised controlled trial. Thorax. 2005 Jun;60(6):480-7. doi: 10.1136/thx.2004.034280. PMID 15923248
- [Background] Donaldson GC, Seemungal T, Jeffries DJ, Wedzicha JA. Effect of temperature on lung function and symptoms in chronic obstructive pulmonary disease. Eur Respir J. 1999 Apr;13(4):844-9. doi: 10.1034/j.1399-3003.1999.13d25.x. PMID 10362051
- [Background] Osman IM, Godden DJ, Friend JA, Legge JS, Douglas JG. Quality of life and hospital re-admission in patients with chronic obstructive pulmonary disease. Thorax. 1997 Jan;52(1):67-71. doi: 10.1136/thx.52.1.67. PMID 9039248
- [Background] Ko FW, Ng TK, Li TS, Fok JP, Chan MC, Wu AK, Hui DS. Sputum bacteriology in patients with acute exacerbations of COPD in Hong Kong. Respir Med. 2005 Apr;99(4):454-60. doi: 10.1016/j.rmed.2004.09.011. PMID 15763452
- [Background] Chang CL, Sullivan GD, Karalus NC, Mills GD, McLachlan JD, Hancox RJ. Predicting early mortality in acute exacerbation of chronic obstructive pulmonary disease using the CURB65 score. Respirology. 2011 Jan;16(1):146-51. doi: 10.1111/j.1440-1843.2010.01866.x. PMID 20920140
- [Background] Kiely DG, Cargill RI, Lipworth BJ. Effects of hypercapnia on hemodynamic, inotropic, lusitropic, and electrophysiologic indices in humans. Chest. 1996 May;109(5):1215-21. doi: 10.1378/chest.109.5.1215. PMID 8625670
- [Background] Smith BE, Madigan VM. Non-invasive method for rapid bedside estimation of inotropy: theory and preliminary clinical validation. Br J Anaesth. 2013 Oct;111(4):580-8. doi: 10.1093/bja/aet118. Epub 2013 May 3. PMID 23645929
- See also: Cardiovascular physiology concepts — http://www.cvphysiology.com/Blood%20Pressure/BP014.htm